CLINICAL TRIAL: NCT01882062
Title: Proof of Concept of an Anaplerotic Study Using Brain Phosphorus Magnetic Resonance Spectroscopy in Huntington Disease
Acronym: TRIHEP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C12-62
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2013-12

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Triheptanoin 1g/kg/day (Experimental): All patients received Triheptanoin oil at 1g/kg/day during 1 month
  Interventions: Drug: Triheptanoin 1g/kg/day

INTERVENTIONS:
Drug: Triheptanoin 1g/kg/day

SUMMARY:
The purpose of this project is to study the efficacy of an anaplerotic treatment on brain energy profile evolution at an early stage of the Huntington disease.

ELIGIBILITY:
Inclusion Criteria:

* 5 < UHDRS < 50
* Age > 18 years
* Ability to undergo MR scanning
* Covered by french social security

Exclusion Criteria:

* Evidence of psychiatric disorder
* Attendant neurological disorder
* Contraindications to MRI (claustrophobia, metallic or material implants)
* Severe head injury
* Unable to understand the protocol
* Pregnancy
* Failure to give informed consent
* Subjects with exclusion criteria required by french law (e.g. subjects who require a legally authorized representative to obtain consent)
* Unwillingness to be informed in case of abnormal MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brain and Spine Institute, Paris, France

REFERENCES:
- [Result] Adanyeguh IM, Rinaldi D, Henry PG, Caillet S, Valabregue R, Durr A, Mochel F. Triheptanoin improves brain energy metabolism in patients with Huntington disease. Neurology. 2015 Feb 3;84(5):490-5. doi: 10.1212/WNL.0000000000001214. Epub 2015 Jan 7. PMID 25568297
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/25568297

RESULTS

PARTICIPANT FLOW:
Groups:
- Triheptanoin Oil at 1g/kg/Day for 1 Month: Patients received triheptanoin oil at 1g/kg/day for 1 month
Period: Overall Study
Arm/Group | Triheptanoin Oil at 1g/kg/Day for 1 Month
Started | 10 (16th of may 2013)
Completed | 10 (18th of july 2013)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Triheptanoin Oil at 1g/kg/Day for 1 Month
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Inorganic Phosphate (Pi) Over Phosphocreatine (PCr): Pi/PCr
Description: The Pi/PCr Ratio is a measure of brain metabolism and it is an index of mitochondrial oxidative regulation.
  A 6-cm 31P transmit/receive surface coil (RAPID Biomedical GmbH, Rimpar, Germany) was used to collect free induction decays for 4 minutes at rest, 8 minutes during visual activation with 6-Hz red/black checkerboard flashes, and 8 minutes after stimulation. Subjects were able to focus on the flashes with a nonmagnetic mirror mounted above their eyes while all lights in the room were turned off. The Pi/PCr ratio was then calculated to determine brain response to cortical activation.
Time Frame: visit 1 (baseline), visit 2 (after 1 month of treatment)
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Triheptanoin Oil at 1g/kg/Day for 1 Month: All the participants received triheptanoin oil at 1g/kg/day for 1 month
Arm/Group | Triheptanoin Oil at 1g/kg/Day for 1 Month
Number analyzed (Participants) | 10
ratio
  Pi/PCr - rest at visit#1 | 0.44 (0.09)
  Pi/PCr - visual stimulation at visit#1 | 0.43 (0.04)
  Pi/PCr - recovery at visit#1 | 0.44 (0.08)
  Pi/PCr - rest at visit#2 | 0.42 (0.05)
  Pi/PCr - visual stimulation at visit#2 | 0.45 (0.05)
  Pi/PCr - recovery at visit#2 | 0.42 (0.04)

2. Secondary Outcome: Correlation Between Primary Outcome Measure and Clinical Parameters
Description: Correlating an improvement of brain energy profile with clinical parameters in Huntington patients such as the Unified Huntington's disease rating scale (UHDRS) and total functional capacity score (TFC).
Time Frame: visit 1 (baseline), visit 2 (after 1 month of treatment)
Reporting Status: Not Posted, anticipated posting 2015-12

ADVERSE EVENTS:
Arm/Group | Triheptanoin Oil at 1g/kg/Day for 1 Month
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No